CLINICAL TRIAL: NCT06187025
Title: Addiction in the Secondary Prevention of Stroke
Brief Title: Addiction & Stroke
Acronym: ADDICT-STROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/56
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Transient Ischemic Attack; Substance Related and Addiction Disorders; Mood disorders; Anxiety Disorders; Secondary prevention
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Mood Disorders; Anxiety Disorders | interventions — Ethanol; Smoking Devices; Insemination, Artificial, Heterologous; Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized clinical evaluations, and screening of substance use (Other): Standardized clinical evaluations, and screening of substance use will be performed for all using the World Health Organization Alcohol, Smoking and Drug Abuse Screening Test (ASSIST).
  Interventions: Other: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST); Other: Ecological Momentary Assessment (EMA)

INTERVENTIONS:
Other: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) — Standardized clinical evaluations and screening of substance use using the World Health Organization Alcohol, Smoking and Drug Abuse Screening Test (ASSIST)
Other: Ecological Momentary Assessment (EMA) — Daily EMA evaluations during 12 weeks

SUMMARY:
Modifiable stroke risk-factors, which include poor lifestyle habits, account for 90 % of the risk of stroke. Disability Adjusted Life Years (DALYs) related to cerebrovascular disorders rely on three main factors, including the severity of stroke-related symptoms, the occurrence of stroke complications, and stroke recurrences.

Stroke complications and the risk of stroke recurrence are highly dependent on the control of vascular risk factors. Thus, the secondary prevention of stroke involves profound lifestyle modifications including substance use cessation and diet changes.

DETAILED DESCRIPTION:
National guidelines for stroke clinical practice advocate an immediate cessation of consumption of all substances but without recommendations on specific therapeutic regimens. Yet, the ability to engage and maintain such lifestyle changes depend on the patient's mental health status. Moreover, independently of stroke, emotional impairments or disorders and substance related and addiction disorders (SRADs) are frequent comorbid conditions (dual disorders) with debilitating consequences and the interplay between the two conditions makes rehabilitation more complex.

Post-stroke emotional impairments are frequent, post-stroke depression and anxiety being the most frequent with a prevalence of 30% and 25% respectively. The consequences of these "invisible handicaps" are observable across a wide range of stroke clinical outcomes. They have been shown to be associated with increased mortality, reduced functional status, decreased quality of life, medication adherence, efficient use of rehabilitation services and cognitive impairment.

Conversely, despite the obvious connection between drugs and stroke, the prevalence and types of SRADs among stroke patients together with their impact and potential interplay with emotional impairments on post-stroke outcomes are still overlooked. The literature is too sparse to guide clinical practice.

Paradoxically, clinicians are facing the devastating effects of addiction in this population and must be informed by solid empirical data. Moreover, the COVID19 pandemic has critically favored or exacerbated poor lifestyle habits (legal and illicit drug use, compulsive overeating) and negative affectivity - including mood and anxiety disorders -, not only in the adult but also the adolescent population. In this context, we believe it is legitimate to expect a noticeable impact on stroke incidence and prognosis in the coming years.

It thus appears that there is an urgent need to allow stroke healthcare professionals to be better equipped to screen and treat problematic substance use in stroke patients. The WHO promotes tools that could effectively support these two priorities.

First, the WHO sponsored the development of the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) to address the need for a reliable and valid screening test. The core criteria chosen for the development of such an instrument were the following: adaptable to different cultures, languages and settings; flexible enough to identify different substances and different patterns of substance use; capable of screening for risk as well as for confirmed cases; ability to link easily into a brief intervention; available at a reasonable/or no cost. Planning and development of the instrument followed a three-phase program; the instrument that is currently available is the ASSIST version 3, for which the French language validation has been already conducted among clients attending primary health care, psychiatric, addiction, and geriatric treatment facilities. These study findings strongly suggest that the ASSIST tool would be suitable for stroke populations.

Additionally, the potential pivotal role of eHealth development has been advocated by the WHO, who considers e-health as a cost-effective and secure use of information and communication technologies (ICT) in support of health and health-related fields. There is a pressing need to develop such a device for the early detection of post-stroke neuropsychiatric complications for each individual patient. The rapid expansion of ambulatory monitoring techniques, such as Ecological Momentary Assessment (EMA), allows daily evaluations of symptoms in real time and in the natural contexts of daily life. We have previously validated the feasibility and validity of EMA to assess daily life emotional symptoms after stroke, demonstrating its utility to investigate their evolution during the 3 months following stroke and to identify early predictors of post-stroke depression such as stress reactivity and social support, suggesting that EMA could be used in the early personalized care management of these neuropsychiatric complications. Moreover, we have developed an Ecological Momentary Intervention via smartphone to improve the outcome of post-stroke emotional status. This eHealth device uses algorithms for detecting at-risk patients depending on the level of mood symptomatology (DSM5 criteria for depression, generalized anxiety, post-traumatic stress disorder, suicidal risk) measured by a daily 3-5 min EMA at the end of the day. Data are sent on-line via secured servers and coded alerts are sent to the hospital clinical team in case risk levels are reached and/or if high levels of symptom persist. This approach permits clinicians to rapidly contact patients and to initiate psychiatric care without requiring the usual 4-month wait (on average) before the standard care follow-up visit. Specifically, based on the alerts, the care pathway is adapted according to each individual condition. The eHealth device is flexible and can be optimized by implementing algorithms and alerts indexing difficulties in controlling substance and unhealthy food intake.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years of age and younger than 80 years;
* Recent (≤ 15 days) clinically symptomatic ischemic or hemorrhagic stroke documented through brain imaging (CT or MRI) or a Transient Ischemic Attack with an ABCD2 score ≥ 4;
* Returning to the Bordeaux Hospital neurovascular unit for the standard care 3-months post-stroke follow-up visit;
* National Institute Health Stroke Scale (NIHSS) < 15;
* modified Rankin scale ≤ 4;
* No severe cognitive impairment as defined by the neurologist;
* Written informed consent by the patient;
* Coverage by the French National Health Insurance.

For the feasibility study assessing the acceptability of the eHealth device to optimize stroke secondary prevention, additional inclusion criteria will be the ability to use a smartphone and living in an area with internet coverage.

Exclusion Criteria:

* Subarachnoid hemorrhage; Dementia syndrome or other neurologic disorder;
* Severe aphasia (NIHSS item 9 ≥ 2) and/or Severe visual impairment interfering with the completion of evaluations;
* Severely impaired physical and/or mental health that, according to the neurologist, may affect the participant's capacity to participate in the study;
* Pregnancy or breastfeeding;
* Inability to read French;
* Individuals under legal protection or unable to personally express their consent
* Participation in another protocol modifying the patient's follow-up status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Organization Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Day 0
  8 questions covering tobacco, alcohol, cannabis, amphetamine type stimulants, inhalants, sedatives, hallucinogens, opiates and 'other drugs' (e.g. sugar, caffeine; fatty food items will be included). It begins by a screening item that asks about lifetime use. In case of a " No " answer, the evaluation terminates. When a " Yes " answer is provided, the remaining questions ask for the substances endorsed during the prior 3 months: 1) the frequency of use, 2) problems and usage patterns, 3) the compulsion to use (psychological dependence), 4) the domains of the problems (personal, health, financial, legal), 5) failure in meeting role obligations, 6) a screening of lifetime in addition to recent problems, 7) attempts at controlling substance use, and 8) current and lifetime injection of drugs (if appropriate). Twenty-eight domains/scores are derived from these questions
Organization Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | 12 Month
  8 questions covering tobacco, alcohol, cannabis, amphetamine type stimulants, inhalants, sedatives, hallucinogens, opiates and 'other drugs' (e.g. sugar, caffeine; fatty food items will be included). It begins by a screening item that asks about lifetime use. In case of a " No " answer, the evaluation terminates. When a " Yes " answer is provided, the remaining questions ask for the substances endorsed during the prior 3 months: 1) the frequency of use, 2) problems and usage patterns, 3) the compulsion to use (psychological dependence), 4) the domains of the problems (personal, health, financial, legal), 5) failure in meeting role obligations, 6) a screening of lifetime in addition to recent problems, 7) attempts at controlling substance use, and 8) current and lifetime injection of drugs (if appropriate). Twenty-eight domains/scores are derived from these questions
Addiction Severity Index - Lite version (ASI) | Day 0
  shortened version of the Addiction Severity Index (French version Denis et al., 2016). It covers areas that may be affected by addiction: medical status, employment/support status, drug and alcohol use, family and social relationships, legal and psychological status. It provides lifetime information as well as over the previous 30 days
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | Day 0
  abbreviated, 13-item version of the Yale Food Addiction Scale 2.0 (mYFAS 2.0; French version Brunault et al., 2020), which was designed specifically to assess signs of addictive-like eating behavior. It includes one question to assess each of the 11 DSM 5 diagnostic criteria for SRADs with two questions to assess clinically significant distress and impairment. There are two scoring options: 1) a "symptom count" that reflects the number of addiction-like criteria endorsed and 2) a "diagnosis" when the participant endorses 2 or more symptom criteria plus clinically significant impairment or distress). FA is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress. It will be proposed either as a self-report or an interviewer-based questionnaire as decided by the psychologist
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | 12 Month
  abbreviated, 13-item version of the Yale Food Addiction Scale 2.0 (mYFAS 2.0; French version Brunault et al., 2020), which was designed specifically to assess signs of addictive-like eating behavior. It includes one question to assess each of the 11 DSM 5 diagnostic criteria for SRADs with two questions to assess clinically significant distress and impairment. There are two scoring options: 1) a "symptom count" that reflects the number of addiction-like criteria endorsed and 2) a "diagnosis" when the participant endorses 2 or more symptom criteria plus clinically significant impairment or distress). FA is mild if there are 2 or 3 symptoms and clinically significant impairment/distress, moderate if there are 4 or 5 symptoms and significant impairment/distress, and severe if there are 6 or more symptoms and significant impairment/distress. It will be proposed either as a self-report or an interviewer-based questionnaire as decided by the psychologist
Fagerström Test for Nicotine Dependence (FTND) Score | Day 0
  includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity
Fagerström Test for Nicotine Dependence (FTND) Score | 3 Month
  includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity
Fagerström Test for Nicotine Dependence (FTND) Score | 6 Month
  includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity
Fagerström Test for Nicotine Dependence (FTND) Score | 12 Month
  includes 10 items. Scores can range from 0 to 10. The recommended cut-off scores to index the categories of nicotine dependence severity are as follows: below 2 = no dependence, 3 to 4 = mild severity, 5 to 6 = moderate severity, 7 to 10 = extreme severity
Alcohol Use Disorder Identification Test (AUDIT) Score | Day 0
  includes 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, above 12 = extreme severity for both sexes
Alcohol Use Disorder Identification Test (AUDIT) Score | 3 Month
  includes 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, above 12 = extreme severity for both sexes
Alcohol Use Disorder Identification Test (AUDIT) Score | 6 Month
  includes 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, above 12 = extreme severity for both sexes
Alcohol Use Disorder Identification Test (AUDIT) Score | 12 Month
  includes 10 items. Scores can range from 0 to 40. The recommended cut-off scores to index the categories of alcohol dependence severity are as follows: from 6 to 12 for women and 7 to 12 for men = moderate severity, above 12 = extreme severity for both sexes
Cannabis Abuse Screening Test (CAST) Score | Day 0
  includes 6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, 3 or more = high risk of dependence
Cannabis Abuse Screening Test (CAST) Score | 3 Month
  includes 6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, 3 or more = high risk of dependence
Cannabis Abuse Screening Test (CAST) Score | 6 Month
  includes 6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, 3 or more = high risk of dependence
Cannabis Abuse Screening Test (CAST) Score | 12 Month
  includes 6 items. Scores can range from 0 to 6. The recommended cut-off scores to index the categories of cannabis dependence severity are as follows: below 2 = low risk of dependence, a score of 2 = moderate risk of dependence, 3 or more = high risk of dependence
Readiness Ruler or Substance Use Motivation Ruler Score | Day 0
  asks the respondent to rank his/her motivation to end his/her substance use on a VAS scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations
Readiness Ruler or Substance Use Motivation Ruler Score | 3 Month
  asks the respondent to rank his/her motivation to end his/her substance use on a VAS scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations
Readiness Ruler or Substance Use Motivation Ruler Score | 6 Month
  asks the respondent to rank his/her motivation to end his/her substance use on a VAS scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations
Readiness Ruler or Substance Use Motivation Ruler Score | 12 Month
  asks the respondent to rank his/her motivation to end his/her substance use on a VAS scale from 1 (Absolutely no motivation to quit) to 10 (No doubt about the decision to be sober) and to list some motivations
Multidimensional Assessment of Thymic States scale (MAThYS) | Day 0
  evaluation of a broad spectrum of mixed mood states. It is based on the concept that mood can be defined using emotional reactivity and not only tonality of affects. It consists in a visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped in five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. motivation and 5. sensory perception.
Multidimensional Assessment of Thymic States scale (MAThYS) | 3 Month
  evaluation of a broad spectrum of mixed mood states. It is based on the concept that mood can be defined using emotional reactivity and not only tonality of affects. It consists in a visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped in five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. motivation and 5. sensory perception.
Multidimensional Assessment of Thymic States scale (MAThYS) | 6 Month
  evaluation of a broad spectrum of mixed mood states. It is based on the concept that mood can be defined using emotional reactivity and not only tonality of affects. It consists in a visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped in five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. motivation and 5. sensory perception.
Multidimensional Assessment of Thymic States scale (MAThYS) | 12 Month
  evaluation of a broad spectrum of mixed mood states. It is based on the concept that mood can be defined using emotional reactivity and not only tonality of affects. It consists in a visual analog scale of 20 items relating to individual states as perceived by the patient for the preceding week. Items can be grouped in five quantitative dimensions ranging each from inhibition to excitation: 1. emotional reactivity, 2. thought processes, 3. psychomotor function, 4. motivation and 5. sensory perception.
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) Score | Day 0
  standardized instrument that has been developed to quickly evaluate post-stroke cognitive, emotional and behavioral complaints. It includes 13 cognitive items, 9 emotional items and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. Scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) Score | 3 Month
  standardized instrument that has been developed to quickly evaluate post-stroke cognitive, emotional and behavioral complaints. It includes 13 cognitive items, 9 emotional items and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. Scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) Score | 6 Month
  standardized instrument that has been developed to quickly evaluate post-stroke cognitive, emotional and behavioral complaints. It includes 13 cognitive items, 9 emotional items and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. Scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
Checklist for Cognitive and Emotional Consequences following stroke (CLCE-24) Score | 12 Month
  standardized instrument that has been developed to quickly evaluate post-stroke cognitive, emotional and behavioral complaints. It includes 13 cognitive items, 9 emotional items and 2 additional open-ended, non-specified items concerning potential additional difficulties not evaluated by the other items. Scoring of each item ranges from 0 (not present) to 3 (present and affecting daily life).
EuroQoL 5-Dimensions Questionnaire (EQ-5D) | 3 Month
  standardized instrument for use as a measure of health outcome in stroke and was designed for self-completion by respondents. The 5 items of the questionnaire provide a simple descriptive profile and a single index value for health status. The EQ-Index has shown reasonable validity and acceptable responsiveness for detecting the health-related quality of life in stroke patients (Chen et al., 2016). This questionnaire has been used in several stroke studies and is currently the primary outcome measure of the Stroke and Carer Optimal Health Program trial
EuroQoL 5-Dimensions Questionnaire (EQ-5D) | 6 Month
  standardized instrument for use as a measure of health outcome in stroke and was designed for self-completion by respondents. The 5 items of the questionnaire provide a simple descriptive profile and a single index value for health status. The EQ-Index has shown reasonable validity and acceptable responsiveness for detecting the health-related quality of life in stroke patients (Chen et al., 2016). This questionnaire has been used in several stroke studies and is currently the primary outcome measure of the Stroke and Carer Optimal Health Program trial
Stroke Risk | Day 0
  The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction
Stroke Risk | 3 Month
  The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction
Stroke Risk | 6 Month
  The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction
Stroke Risk | 12 Month
  The Stroke Riskometer app assesses the possibility of suffering a stroke using a number of health and lifestyle factors including age, sex, ethnic origin, blood pressure, atrial fibrillation, left ventricular hypertrophy, anti-hypertension, tobacco, cardiovascular history, weight / height ratio, cholesterol level, diabetes, alcohol, stress, cognitive decline, family and personal history of stroke and TIA, history of head trauma and myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Igor Sibon, Principal Investigator — University Hospital, Bordeaux; Sylvie Berthoz, Study Director — CNRS UMR 5287 - INCIA
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No